CLINICAL TRIAL: NCT01459497
Title: Phase III Randomized Study of Standard Versus Accelerated Hypofractionated Image-Guided Radiation Therapy (IGRT) in Patients With Stage II-III Non-Small Cell Lung Cancer and Poor Performance Status
Brief Title: Hypofractionated Image-Guided Radiation Therapy (IGRT) in Patients With Stage II-III Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Puneeth Iyengar, Associate Vice Chair of Clinical Research, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU 052011-093
Record Dates: First submitted 2011-10-19; First posted 2011-10-25 (Estimated); Results first posted 2022-05-16 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Non-small Cell Lung Cancer
Keywords: non-small cell lung cancer; Stages II or III non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Radiation Therapy (Active Comparator): Arm A:Image-Guided Radiation Therapy (IGRT), 60 Gy in 15 fractions in 3 weeks
  Interventions: Radiation: Radiation Therapy
- Conventional Radiation (Active Comparator): Arm B: Conventional radiation 60-66 Gy in 30-33 fractions in 6-7 weeks
  Interventions: Radiation: Conventional radiation

INTERVENTIONS:
Radiation: Radiation Therapy — Image-Guided Radiation Therapy (IGRT)60 Gy in 15 fractions in 3 weeks
  Arms: Radiation Therapy
Radiation: Conventional radiation — Conventional radiation 60-66 Gy in 30-33 fractions in 6-7 weeks
  Arms: Conventional Radiation

SUMMARY:
The study is designed to determine whether an accelerated course of hypofractionated radiation therapy with daily image guidance and motion assessment/control will allow more effective treatment of poor performance status patients with stage II-III NSCLC, who would benefit from local therapy compared to standard radiation therapy (60 Gy in 2 Gy per fraction).

DETAILED DESCRIPTION:
The study is designed to determine whether an accelerated course of hypofractionated radiation therapy with daily image guidance and motion assessment/control will allow more effective treatment of poor performance status patients with stage II-III NSCLC, who would benefit from local therapy compared to standard radiation therapy (60 Gy in 2 Gy per fraction). Poor performance status patients can be a heterogeneous group, with tumor-related factors, other co-morbidities, or advanced age placing patients in the category. These patients have traditionally been underrepresented in clinical trials, and thus no prospective study has evaluated the efficacy of other radiotherapy dose fractionations in these patients. One phase III trial of "poor-risk" locally advanced NSCLC (RTOG 93-04) included just over 40% Karnofsky performance status 60-70 patients and showed median survival times of 9.5 and 10.3 months with 60Gy of conventional radiation therapy alone or with recombinant β-interferon [18]. 1 year overall survival was just 44% in these patients.

This study includes randomization to two arms. Arm A (experimental arm) will include IGRT, 60 Gy in 15 fractions (3 weeks). Arm B will include conventional radiation, 60-66 Gy in 30-33 fractions (6 weeks) with optional concurrent with carboplatin/taxol .

The experimental arm dose for this trial is based on a dose escalation trial at University of Texas Southwestern evaluating the maximum tolerated dose of hypofractionated IGRT in this patient population (Phase I study IRB #072010-050). Doses were escalated from 3 Gy per fraction (total dose 45 Gy) to 4 Gy per fraction (total dose 60 Gy) and evaluation for treatment related toxicity was being performed. Critical structure dose constraints will be expressed as organ dose-volume limits, with limits formulated with the approval of the study investigators using known tolerance data, radiobiological conversion models, and norms used in current practice at academic centers [27].

Randomization Schema:

Patients will be allocated to the treatment using a randomized permuted block within strata to balance for patient factors other than institution. The stratifying variables are Zubrod performance status (2 vs. > 2) and stage (II vs. III).

ELIGIBILITY:
Inclusion Criteria:

* All patients must be willing and capable to provide informed consent to participate in the protocol.
* Patients must have appropriate staging studies identifying them as AJCC stage II or III non small cell lung cancer, (according to AJCC Staging, 6th edition; see appendix III), or recurrent non small cell lung cancer. Histologic confirmation of cancer will be required by biopsy or cytology within 6 months of study entry.
* Patients must have the potential for benefit from local therapy (at the discretion of the investigator).
* The patient's Zubrod performance status must be 2 or greater OR patients with Zubrod performance status 0-1 and weight loss >10% are considered eligible. In addition, patients determined to be medically unfit or refusing combined modality therapy are eligible.
* Age ≥ 18.
* Patients must have measurable or evaluable disease.
* Women of childbearing potential and male participants must agree to use an effective method of contraception.
* Patients must sign study specific informed consent prior to study entry.
* Patients must not have plans for concurrent chemoradiation therapy.
* Patients must complete all required pretreatment evaluations

Exclusion Criteria:

* Total (aggregate) gross tumor volume > 500 cm3 (500 cc's or 0.5 Liters)
* Prior radiotherapy to the region of the study cancer that would result in direct overlap of radiation therapy fields.
* Chemotherapy given within one week of study registration.
* Pregnant or lactating women, as treatment involves unforeseeable risks to the embryo or fetus.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2019-07-11 (Actual); Study Completion 2023-10-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Puneeth Iyengar, MD, Principal Investigator — University of Texas Southwestern Medical Center; Puneeth Iyengar, MD, Principal Investigator — puneeth.iyengar@utsouthwestern.edu
Locations (7):
- United States (7):
  - Georgetown Cancer Center (Austin Cancer Center), Austin, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Md Anderson Cancer Center, Houston, Texas
  - Baylor Research Institute Dallas, Baylor Irving, Irving, Texas
  - Texas Oncology - Sherman, Sherman, Texas
  - Scott & White Memorial Temple, Temple, Texas
  - Texas Oncology - Tyler, Tyler, Texas

REFERENCES:
- [Derived] Iyengar P, Zhang-Velten E, Court L, Westover K, Yan Y, Lin MH, Xiong Z, Patel M, Rivera D, Chang J, Saunders M, Shivnani A, Lee A, Hughes R, Gerber D, Dowell J, Gao A, Heinzerling J, Li Y, Ahn C, Choy H, Timmerman R. Accelerated Hypofractionated Image-Guided vs Conventional Radiotherapy for Patients With Stage II/III Non-Small Cell Lung Cancer and Poor Performance Status: A Randomized Clinical Trial. JAMA Oncol. 2021 Oct 1;7(10):1497-1505. doi: 10.1001/jamaoncol.2021.3186. PMID 34383006

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Radiation Therapy | Conventional Radiation
Started | 52 | 51
Completed | 50 | 46
Not Completed | 2 | 5
Not completed — Inability to meet trial constraints. | 1 | 0
Not completed — Physician Decision | 1 | 1
Not completed — Hospitalization. | 0 | 3
Not completed — Disease progression. | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Radiation Therapy | Conventional Radiation | Total
Number analyzed (Participants) | 50 | 46 | 96
Age, Customized [Count of Participants; unit: Participants]
  Ages 50-59 years | 6 | 9 | 15
  Ages 60-69 years | 13 | 12 | 25
  Ages 70-79 years | 18 | 17 | 35
  Ages 80-90 years | 13 | 8 | 21
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 13 | 33
  Male | 30 | 33 | 63
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 31 | 30 | 61
  Black | 18 | 16 | 34
  Asian | 1 | 0 | 1
Region of Enrollment [Number; unit: number of participants]
  United States | 50 | 46 | 96
Baseline performance status [Count of Participants; unit: Participants] — Zubrod Performance Scale will be used:
  0 Fully active, able to carry on all predisease activities without restriction;
  1. Restricted in physically strenuous activity but ambulatory and able to carry work of a light or sedentary nature. For example, light housework, office work;
  2. Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours;
  3. Capable of only limited self-care, confined to bed or chair 50% or more of waking hours;
  4. Completely disabled. Cannot carry on self-care. Totally confined to bed;
  5. Death
  Participants
    0 | 1 | 1 | 2
    1 | 16 | 13 | 29
    2 | 28 | 29 | 57
    3 | 5 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival of Standard Radiation (CFRT) Versus Accelerated, Hypofractionated, Image-guided Conformal Radiotherapy (IGRT) in Treatment of Stage II-III NSCLC in Patients With Poor Performance Status at 1 Year.
Description: Percentage of participants with overall survival at 1 year. To compare the efficacy by overall survival of standard radiation versus accelerated, hypofractionated, image-guided conformal radiotherapy in treatment of stage II-III or recurrent NSCLC in patients with poor performance status. Overall survival time will be estimated using the Kaplan-Meier approach. The stratified log-rank test will be used to test for a statistically significant difference in survival distributions. The Cox proportional hazard regression model will be used to determine hazard ratios and 95% confidence intervals for the treatment difference in overall survival. Unadjusted ratios and ratios adjusted for stratification variables and other covariates of interest will be computed.
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Radiation Therapy | Conventional Radiation
Number analyzed (Participants) | 50 | 46
percentage of participants | 37.7 [24.2 to 51.0] | 44.6 [29.9 to 58.3]

2. Secondary Outcome: Toxicities of Two Radiotherapy Treatment Regimens in Patients With Stage II-III Non-Small Cell Lung Cancer (NSCLC) and Poor Performance Status
Description: To compare toxicity of two radiotherapy treatment regimens in patient with stage II-III Non-Small Cell Lung Cancer (NSCLC) and poor performance status. Toxicity will be assessed according to the NCI Common Toxicity Criteria for Adverse Events (CTCAE), version 4.0.
Time Frame: 60 months
Measure: Number; unit: events
Arm/Group | Radiation Therapy | Conventional Radiation
Number analyzed (Participants) | 50 | 46
events | 144 | 120

3. Secondary Outcome: Time to Local Progression of Two Radiotherapy Treatment Regimens in Patients With Stage II-III NSCLC and Poor Performance Status
Description: The time to disease progression and time to local regression will be estimated using the Kaplan-Meier approach. The stratified log-rank test will be used to test for a statistically significant difference in PFS (progression-free survival) and time to local progression distributions. The Cox proportional hazard regression model will be used to determine hazard ratios and 95% confidence intervals for the treatment difference in progression-free survival and time to local progression. Time to progression will be measured from the date of study enrollment to the date of documented local progression as determined by clinical exam and imaging studies.
Time Frame: 60 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Radiation Therapy | Conventional Radiation
Number analyzed (Participants) | 50 | 46
months | 6.4 [4.1 to 7.8] | 7.3 [5.0 to 10.6]

4. Secondary Outcome: Disease-free Survival of Two Radiotherapy Treatment Regimens in Patients With Stage II-III NSCLC and Poor Performance Status.
Description: Percentage of patients with disease-free survival at 60 months. To compare disease-free survival of two radiotherapy treatment regimens in patients with stage II-III NSCLC and poor performance status. Unlike progression-free survival in the advanced cancer setting, which refers to time from treatment to disease progression (or death) in patients who already have measurable cancer in their bodies, DFS (disease-free survival) refers to time from treatment until the recurrence of disease (or death) after undergoing curative-intent treatment.
Time Frame: 60 months
Measure: Number; unit: percentage of participants
Arm/Group | Radiation Therapy | Conventional Radiation
Number analyzed (Participants) | 50 | 46
percentage of participants | 4 | 2

5. Secondary Outcome: Quality of Life of Two Radiotherapy Treatment Regimens in Patients With Stage II-III NSCLC and Poor Performance Status.
Description: Patient-reported functional status will be assessed with the lung cancer subscales of the Functional Assessment of Cancer Therapy-Lung (FACT-L). The FACT-L is a 36-item questionnaire that uses 5-point Likert-type response choices (0 = not at all; 1 = a little bit; 2 =somewhat; 3 = quite a bit; 4 = very much).
Time Frame: 6 months
Population: Data was not collected due to patient compliance.
Arm/Group | Radiation Therapy | Conventional Radiation
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Cost Effectiveness of Two Radiotherapy Treatment Regimens in Patients With Stage II-III NSCLC and Poor Performance Status.
Description: For the primary analysis, we will estimate cost accumulated within 2 years. An inverse-probability weighting method to calculate average costs for each treatment group will be used to analyze.
Time Frame: 2 years
Population: Due to patient compliance with questionnaire completion, only 23 patients from Arm A and 29 patients from Arm B were analyzed. Sample size was too small for meaningful cost comparison.
Measure: Mean (95% Confidence Interval); unit: Cost of Treatment (in USD)
Arm/Group | Radiation Therapy | Conventional Radiation
Number analyzed (Participants) | 23 | 29
Cost of Treatment (in USD) | 26,984 [14714 to 39253] | 33,723 [12188 to 55256]

7. Secondary Outcome: Quality Adjusted Life Survival Time of Two Radiotherapy Treatment Regimens in Patients With Stage II-III NSCLC and Poor Performance Status.
Description: The quality-adjusted survival time is just an integration of the utility measures over a patient's survival time, or until the time limit similar as the cost calculation, whichever occurs earlier. To estimate quality adjusted survival time, data from EQ-5D (EuroQol- 5 Dimension a descriptive system for health-related quality of life states in adults), each of which has five severity levels that are described by statements appropriate to that dimension) will first be translated into utility measures. These measures are obtained at discrete time points, so they will be interpolated into the time intervals between the visits. Accordingly, we will use the inverse-probability weighted method of Zhao and Tsiatis to carry out the survival time analysis.
Time Frame: 20 months
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Radiation Therapy | Conventional Radiation
Number analyzed (Participants) | 23 | 29
days | 100 [70 to 130] | 81 [48 to 115]

8. Secondary Outcome: Quality Adjusted Life Survival Time of Two Radiotherapy Treatment Regimens in Patients With Stage II-III NSCLC and Poor Performance Status.
Description: The quality-adjusted survival time is just an integration of the utility measures over a patient's survival time, or until the time limit similar as the cost calculation, whichever occurs earlier. To estimate quality adjusted survival time, data from the VAS (visual analogue scale: the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine') of EQ-5D (EuroQol- 5 Dimension a descriptive system for health-related quality of life states in adults), each of which has five severity levels that are described by statements appropriate to that dimension) will first be translated into utility measures. These measures are obtained at discrete time points, so they will be interpolated into the time intervals between the visits. Accordingly, we will use the inverse-probability weighted method of Zhao and Tsiatis to carry out the survival time analysis.
Time Frame: 20 months
Measure: Mean (95% Confidence Interval); unit: adjusted days of follow up
Arm/Group | Radiation Therapy | Conventional Radiation
Number analyzed (Participants) | 23 | 29
adjusted days of follow up | 106 [73 to 139] | 83 [45 to 122]

ADVERSE EVENTS:
Time Frame: 60 months
Description: Adverse events will be graded by a numerical score according to the defined NCI Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 4.0: Grade 1: Mild; Grade 2: Moderate; Grade 3: Severe or medically significant but not immediately life threatening; Grade 4: Life threatening consequences; Grade 5: Death related to the adverse event
Arm/Group | Radiation Therapy | Conventional Radiation
All-Cause Mortality (participants affected / at risk) | 32/50 | 26/46
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/46
Other Adverse Events (participants affected / at risk) | 28/50 | 23/46
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiation Therapy (N=50) | Conventional Radiation (N=46)
Pericardial Effusion (Cardiac disorders) | 0 (0) | 1 (1)
SVC (Superior vena cava) Syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Fatigue (Nervous system disorders) | 23 (23) | 23 (23)
Anorexia (Gastrointestinal disorders) | 7 (7) | 10 (10)
Dysphagia (Gastrointestinal disorders) | 12 (12) | 10 (10)
Esophagitis (Gastrointestinal disorders) | 20 (20) | 16 (16)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chest Wall Pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3)
ARDS (Acute respiratory distress syndrome) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 11 (11)
DLCO (Diffusion capacity of carbon monoxide) decline (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 28 (28) | 13 (13)
FEV (forced expiratory volume) decline (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 5 (5)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 8 (8) | 6 (6)
Dryness (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Our study has several limitations. First, it was closed to accrual before the enrollment goal was attained due to futility in reaching the primary endpoint; consequently, the lower than anticipated number of participants limited our multivariate analysis. Second, more than half of the patients were from a single site (University of Texas Southwestern). Finally, the outcomes may have differed in an immuno-therapy setting.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-05-22): https://cdn.clinicaltrials.gov/large-docs/97/NCT01459497/Prot_SAP_ICF_000.pdf